CLINICAL TRIAL: NCT01578720
Title: Treatment of CNV Secondary to Presumed Ocular Histoplasmosis With EYLEA 2.0mg (Intravitreal Aflibercept Injection)
Brief Title: Intravitreal Aflibercept Injection (IAI) for Presumed Ocular Histoplasmosis Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Retina Research Institute, LLC (Other)
Responsible Party: Principal Investigator, Rhonda Weeks, Kevin J. Blinder, MD, Retina Research Institute, LLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KB-001
Record Dates: First submitted 2012-04-02; First posted 2012-04-17 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Choroidal Neovascularization; Presumed Ocular Histoplasmosis
MeSH Terms: conditions — Choroidal Neovascularization | interventions — aflibercept; Intravitreal Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IVT injection once every 8 weeks after 3 initial monthly doses (Other): Intravitreal aflibercept injection 2.0mg dosed every 4 weeks (monthly)for the first 3 months followed by 2.0 mg (0.05mL) via intravitreal injection every eight weeks (2 months).
  Dosing at monthly intervals is allowed if needed in the opinion of the investigator based on presence of fluid on OCT and/or a decrease in visual acuity of greater than or equal to 5 letters from the previous visit.
  Interventions: Drug: EYLEA (Aflibercept) intravitreal injection

INTERVENTIONS:
Drug: EYLEA (Aflibercept) intravitreal injection — Intravitreal Injection once every 8 weeks with 3 initial monthly doses

SUMMARY:
The purpose of this study is to assess the efficacy and safety of intravitreal injection of aflibercept for the treatment of Choroidal Neovascularization (CNV) secondary to presumed ocular histoplasmosis syndrome (POHS).

ELIGIBILITY:
Inclusion Criteria:

* CNV of less than 1 year duration due to presumed ocular histoplasmosis
* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age 21 years and older
* Subfoveal or juxtafoveal CNV lesion of less than 5400um in diameter
* Best corrected visual acuity of 20/25 to 20/400
* Birth control therapy for females of child-bearing age

Exclusion Criteria:

* CNV due to presumed ocular histoplasmosis for greater than 1 year
* Pregnancy (positive pregnancy test) or lactation
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception : surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch
* A recent history of smoking (within 1 year of study enrollment)
* Prior treatment with intravitreal aflibercept injection
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Uncontrolled glaucoma in the study eye (defined as IOP greater or equal to 30 mmHg despite treatment with anti-glaucoma medication)
* History of cerebral vascular accident, myocardial infarction, transient ischemic attacks within 3 months of study enrollment
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Presence of significant subfoveal fibrosis or atrophy
* Intraocular surgery (including cataract surgery) in the study eye within 2 months of enrollment
* Active intraocular inflammation (grade trace or above) in the study eye
* History of allergy to fluorescein, ICG or iodine, not amendable to treatment
* Any concurrent intraocular condition in the study eye (e.g., cataract or diabetic retinopathy) that, in the opinion of the investigator, could either
* Require medical or surgical intervention during the 12 month study period to prevent or treat visual loss that might result from that condition, or
* If allowed to progress untreated, could likely contribute to loss of at least 2 snellen equivalent lines of BCVA over the 12 month study period
* Prior/Concomitant Treatment:
* Panretinal photocoagulation treatment
* Previous intraocular steroids or PDT within 3 months
* Previous participation in any studies of investigational drugs within 30 days preceding Day 0 (excluding vitamins and minerals)
* Previous treatment with intravitreally (in either eye) or intravenously administered Avastin (bevacizumab) within 60 days
* Previous use of Macugen or Lucentis in study eye within 60 days
* Prior submacular or vitreous surgery

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-06; Primary Completion 2014-04 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Safety | 12 months
  The Incidence & Severity will be assessed during study participation. Baseline medical conditions & abnormal findings present prior to the patient signing the Informed Consent Form (ICF)will be recorded as pre-existing illnesses in the medical history. Clinical study staff will start assessing subjects for adverse events once the ICF has been signed starting at month 1 and at each monthly visit,and will be instructed to request the adverse event information in a nonspecific, non-suggestive type of questioning. The Investigators will record all adverse events regardless of causality.

SECONDARY OUTCOMES:
Mean visual acuity (BCVA) at Months 6 and 12 | Month 6 and Month 12
Mean change in OCT central foveal thickness from baseline at Months 6 and 12 | Months 6 and 12
Mean change in Macular Volume from baseline at Months 6 and 12 | Months 6 and 12
Mean change in visual acuity (BCVA) from baseline at Months 6 and 12 | Months 6 and 12
Mean change in CNV lesion characteristics (size, leakage, etc.) from baseline at Months 6 and 12 | Months 6 and 12
Proportion of patients with no fluid on OCT (absence of cystic edema and subretinal fluid) at Months 6 and 12 | Months 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J Blinder, MD, Principal Investigator — The Retina Institute
Locations (1):
- The Retina Institute, St Louis, Missouri, United States